CLINICAL TRIAL: NCT04138940
Title: Modulating Stimuli Intensity to Improve Clinical Outcomes in Aphasia Treatment
Brief Title: Modulating Intensity and Dosage of Aphasia Scripts
Acronym: MIDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Northwestern University (Other); University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Leora Cherney, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00209618; 1R01DC016979-01A1 (NIH)
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Aphasia
Keywords: Stroke; Speech and Language Therapy; Speech and Language Treatment; Communication Disorders; Language Disorders
MeSH Terms: conditions — Aphasia; Stroke; Communication Disorders; Speech; Language Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Distributed, Short Script (Experimental): Participant practices for 1 hour, 2 days a week for 5 weeks using a 5 sentence-long script.
  Interventions: Behavioral: Script Training
- Distributed, Long Script (Experimental): Participant practices for 1 hour, 2 days a week for 5 weeks using a 10 sentence-long script.
  Interventions: Behavioral: Script Training
- Massed, Short Script (Experimental): Participant practices for 1 hour, 5 days a week for 2 weeks using a 5 sentence-long script.
  Interventions: Behavioral: Script Training
- Massed, Long Script (Experimental): Participant practices for 1 hour, 5 days a week for 2 weeks using a 10 sentence-long script.
  Interventions: Behavioral: Script Training

INTERVENTIONS:
Behavioral: Script Training — Participant uses a computer program to practice scripts with a virtual therapist.

SUMMARY:
The purpose of this study is to evaluate how changing conditions of speech-language treatment (namely, amount of repetition and distribution of practice schedule) affects the language outcome of participants with aphasia following a stroke. Using a computer based speech and language therapy program, participants will practice conversational scripts that are either short or long. Participants will practice for either 2 weeks (5 days a week) or for 5 weeks (2 days a week).

DETAILED DESCRIPTION:
Determining the optimal intensity of treatment is essential to the design and implementation of any treatment program for aphasia. Yet, treatment intensity is a complex construct and information on the variables modulating it remain ambiguous and limited. Studies reported in the neuroscience and clinical literature support the need for intensive treatment to induce long-term neuroplastic changes while the cognitive psychology literature suggests that learning is best maintained with distributed schedules. A few studies have looked at dose parameters for single word naming tasks, but there is limited evidence regarding dose parameters for treatments that focus on training the production of larger units, such as sentences or even connected discourse. One approach that is frequently used clinically and has evidence for its efficacy is script training. Little is currently known regarding the optimum dose of script training (i.e., the number of repetitions over time of each sentence within the script) that is required to promote the best outcomes.

This study investigates the effects of modulating stimulus variables, specifically stimulus practice distribution and stimulus repetition. We use a baseline script treatment that has experimental support regarding its efficacy, and that allows the manipulation of these variables. To ensure independence and fidelity, treatment is provided in a controlled computer environment (desktop and tablet). To avoid clinician-related variables such as expertise and personality factors that may influence treatment, sentences are modeled during treatment by an anthropomorphic agent with high visual speech intelligibility and affective expressions.

With regard to "best outcomes", generalization is the ultimate goal of any treatment approach. Therefore, the primary outcome is a generalization measure of conversation. Secondary measures address short-term acquisition, longer-term maintenance, and stimulus and response generalization for assessing gain over baseline, differential effects, and interactions. A mobile-connected wireless wearable laryngeal sensor allows tracking of talk time at home and in the community as a measure of treatment effectiveness and transfer. For privacy, it does not record audio.

Results and computational models of learning (generalization, short-term acquisition, and longer-term maintenance) will contribute new evidence to fill critical gaps in current scientific understanding regarding the effectiveness and clinical application of aphasia treatment approaches. More generally, findings will help to inform clinical practice and treatment of neurologic communication disorders; the virtual clinician guided intervention that the proposal develops has the potential to reduce costly clinician-client time otherwise required for long-term rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with diagnosis of aphasia
* Left-hemisphere stroke
* Aphasia Quotient score between 40-80 on the Western Aphasia Battery-Revised
* At least 6 months post stroke
* Completed at least eighth grade education
* Premorbidly literate in English
* Visual acuity no worse than 20/100 corrected in the better eye
* Auditory acuity no worse than 30 dB HL on pure tone testing, aided in better ear
* Not receiving speech-language therapy at the time of study

Exclusion Criteria:

* Any other neurological condition (other than cerebral vascular disease) that could potentially affect cognition or speech, such as Parkinson's Disease, Alzheimer's Dementia, traumatic brain injury
* Any significant psychiatric history prior to the stroke, such as severe major depression or psychotic disorder requiring hospitalization; subjects with mood disorders who are currently stable on treatment will be considered
* Active substance abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Generalization - Conversation with a communication partner using the lines of the trained script | Change from baseline to immediately post treatment
  Number of correct information units produced during conversation with communication partner (speech-language pathologist) using the lines of the trained script.

SECONDARY OUTCOMES:
Generalization - Conversation with a communication partner about the topic of the trained script | Change from baseline to immediately post treatment
  Number of correct information units produced during conversation with communication partner (speech-language pathologist) about the broad topic of the trained script.
Acquisition of trained script - Accuracy | Change from baseline to immediately post treatment
  Percent accurate words produced on trained script during oral reading probes provided via the computer program.
Acquisition of trained script - Rate | Change from baseline to immediately post treatment
  Rate of production (words per minute) of trained script during oral reading probes provided via the computer program.

OTHER OUTCOMES:
Maintenance - Conversation with a communication partner using the lines of the trained script | Change from baseline to six weeks post treatment.
  Number of correct information units produced during conversation with communication partner (speech-language pathologist) using the lines of the trained script.
Maintenance - Conversation with a communication partner about the topic of the trained script | Change from baseline to six weeks post treatment.
  Number of correct information units produced during conversation with communication partner (speech-language pathologist) about the broad topic of the trained script.
Maintenance of trained script - Accuracy | Change from baseline to six weeks post treatment
  Percent accurate words produced on trained script during oral reading probes provided via the computer program.
Maintenance of trained script - Rate | Change from baseline to six weeks post treatment
  Rate of production (words per minute) of trained script during oral reading probes provided via the computer program.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Cherney, PhD, CCC-SLP, Principal Investigator — Shirley Ryan Abilitylab, Northwestern University
Locations (1):
- Shirley Ryan Abilitylab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Aphasia Research & Treatment — https://www.sralab.org/research/labs/center-aphasia-research-treatment